CLINICAL TRIAL: NCT02094248
Title: A Randomized, Open-label, Placebo-controlled, Multi-center Study to Evaluate Safety and Efficacy of Recombinant Human Thrombopoietin Among Severe Sepsis Patients With Thrombocytopenia
Brief Title: rhTPO in Critical Patients With Thrombocytopenia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jianan Ren, Vice president of General Surgery Department, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPO Study
Record Dates: First submitted 2014-03-17; First posted 2014-03-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2014-06

CONDITIONS: Sepsis; Thrombocytopenia
MeSH Terms: conditions — Sepsis; Thrombocytopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TPO (Experimental): rhTPO（Recombinant Human Thrombopoietin，TPIAO®, Shenyang Sunshine Pharmaceutical Company Limited [SUNSHINE], Shenyang, China）， 15000U/ml, s.c injection
  Interventions: Drug: TPO
- control (Placebo Comparator): Normal saline，1ml/day, s.c injection
  Interventions: Drug: control

INTERVENTIONS:
Drug: TPO — rhTPO（Recombinant Human Thrombopoietin，TPIAO®, Shenyang Sunshine Pharmaceutical Company Limited [SUNSHINE], Shenyang, China）， 15000U/ml, s.c injection
  Arms: TPO
Drug: control — Normal saline，1ml/day, s.c injection
  Arms: control

SUMMARY:
The primary objectives of this study are to assess the impact of rhTPO on mortality among severe sepsis patients with thrombocytopenia, as well as changes of platelet counts and platelet transfusion rates.

DETAILED DESCRIPTION:
Thrombocytopenia is prevalent among critical patients who is admitted to intensive care unit. Researches have shown that thrombocytopenia is associated with mortality among those patients. Currently, no standard therapy exist for critical patients with Thrombocytopenia. In 2012 SSC guideline, platelet transfusion is induced for thrombocytopenia in critical patients for reducing the risk of bleeding. However, indication for platelet transfusion is relatively strict. No early intervention could be done according to this guideline. Previous studies have shown that recombinant human thrombopoietin can reduce severe sepsis with low platelet 28-day mortality in patients with hyperlipidemia, effectively improve peripheral platelet number, reducing the probability of platelet transfusion.The primary objectives of this study are to assess the impact of rhTPO on mortality among severe sepsis patients with thrombocytopenia, as well as changes of platelet counts and platelet transfusion rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients would be include if Diagnosed as sepsis according to ACCP/CCM criteria Platelet counts is less than 50×109/L for 2 continues days Patient or legally authorized representative able to provide informed consent

Exclusion Criteria:

* Subject has had a splenectomy for any reason Subject has an active malignancy who is now under chemotherapy Subject has a known history of bone marrow stem cell disorder Subject is receiving other investigational agents or procedures Subject is currently enrolled in, or has completed within the last 30 days, another investigational device or drug study Subject is pregnant or breast feeding Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and does not have a legally acceptable representative Subject has any kind of disorder that compromises the ability of the subject to comply with study procedures Subject is less than 18 years or more than 85 years of age History of bone marrow, lung, liver, pancreas, or small-bowel transplantation Acute pancreatitis with no established source of infection

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Mortality | 28-day after enrolled

SECONDARY OUTCOMES:
Time to recover to a normal platelet level | 10 days
Occurrence of bleeding event | 10 days
7-day survival rate | 7 days
Number of Participants who survived from thrombocytopenia | 10 days
Occurrence of platelet transfusion | 10 days
Total amount of platelet transfusion | 10 days
Percentage of participants with platelet response | 10 days
  Platelet response was defined as platelet counts 50 x 10^9/L, measured at each study visit up to the end of the study period
Time to platelet response | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Ren, Study Chair — Department of general surgery, Nanjing Jinling hospital
Locations (1):
- Nanjing Jinling Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Wu Q, Ren J, Wang G, Gu G, Hu D, Liu S, Li G, Chen J, Li R, Hong Z, Ren H, Wu X, Li Y, Yao M, Zhao Y, Li J. Evaluating the safety and efficacy of recombinant human thrombopoietin among severe sepsis patients with thrombocytopenia: study protocol for a randomized controlled trial. Trials. 2015 May 19;16:220. doi: 10.1186/s13063-015-0746-6. PMID 25986785